CLINICAL TRIAL: NCT04816214
Title: A Phase III Randomized, Controlled, Open-label, Multicenter, Global Study of Capmatinib in Combination With Osimertinib Versus Platinum - Pemetrexed Based Doublet Chemotherapy in Patients With Locally Advanced or Metastatic NSCLC Harboring EGFR Activating Mutations Who Have Progressed on Prior Generation EGFR-TKI Therapy and Whose Tumors Are T790M Mutation Negative and Harbor MET Amplification (GEOMETRY-E)
Brief Title: Study Evaluating Efficacy and Safety of Capmatinib in Combination With Osimertinib in Adult Subjects With Non-small Cell Lung Cancers as Second Line Therapy
Acronym: GEOMETRY-E
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Novartis decided to terminate the study based on a business consideration and not related with any safety concerns. Randomized part was not initiated
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CINC280L12301; 2020-003677-21 (EudraCT Number)
Record Dates: First submitted 2021-03-22; First posted 2021-03-25 (Actual); Results first posted 2023-10-30 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: INC280; capmatinib; osimertinib; pemetrexed; platinum-based chemotherapy; NSCLC; Non-Small Cell Lung Cancer; Carcinoma; EGFR Mutation; T790M negative; MET amplification; second line therapy; GEOMETRY; GEOMETRY-E
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma | interventions — capmatinib; osimertinib; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Intervention Model Description: The study was terminated early based on Sponsor's decision unrelated to any safety concerns and the randomized part of the study was not initiated
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Run-in part: Capmatinib + Osimertinib (Experimental): In the run-in part, up to two dose levels of capmatinib in combination with osimertinib were planned to be investigated. The initial dose level for the combination therapy was capmatinib 400 mg orally twice daily (b.i.d) and osimertinib 80 mg orally once per day (q.d). If a dose de-escalation was necessary, a lower dose level was defined as capmatinib 400 mg orally b.i.d and osimertinib 40 mg orally q.d.
  Interventions: Drug: Capmatinib; Drug: Osimertinib
- Randomized part: Capmatinib + Osimertinib (Experimental): In the randomized part, capmatinib in combination with osimertinib was to be administered at the recommended Phase III regimen (defined in the safety run-in part).
  The study was terminated early based on Sponsor's decision unrelated to safety concerns and the randomized part of the study was not initiated.
  Interventions: Drug: Capmatinib; Drug: Osimertinib
- Randomized Part: Platinum + Pemetrexed Based Doublet Chemotherapy (Active Comparator): In the randomized part, platinum-pemetrexed based doublet chemotherapy was to follow local guidelines as per standard of care and products labels. Participants randomized to platinum-pemetrexed based doublet chemotherapy arm were to be allowed to crossover to receive capmatinib in combination with osimertinib. The study was terminated early based on Sponsor's decision unrelated to safety concerns and the randomized part of the study was not initiated.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: Capmatinib — Capmatinib was available as a film-coated tablet for oral use, with a strength of either 150 mg or 200 mg. The initial dose of the combination therapy consisted of capmatinib 400 mg administered orally twice daily (b.i.d).
  Other Names: INC280
  Arms: Randomized part: Capmatinib + Osimertinib; Run-in part: Capmatinib + Osimertinib
Drug: Osimertinib — Osimertinib was available as a tablet for oral use, with a strength of either 80 mg or 40 mg. The initial dose of the combination therapy consisted of osimertinib 80 mg administered orally once per day (q.d)
  Arms: Randomized part: Capmatinib + Osimertinib; Run-in part: Capmatinib + Osimertinib
Drug: Pemetrexed — Pemetrexed concentrate for solution for intravenous use was to be administered intravenously. The procurement of pemetrexed was to be done locally, following local practices and regulations.
  Arms: Randomized Part: Platinum + Pemetrexed Based Doublet Chemotherapy
Drug: Cisplatin — Cisplatin concentrate for solution for intravenous use was to beadministered intravenously during the study. The procurement of cisplatin was to be done locally, following local practices and regulations.
  Arms: Randomized Part: Platinum + Pemetrexed Based Doublet Chemotherapy
Drug: Carboplatin — Carboplatin concentrate for solution for intravenous use was to be administered intravenously during the study. The procurement of carboplatin was to be done locally, following local practices and regulations.
  Arms: Randomized Part: Platinum + Pemetrexed Based Doublet Chemotherapy

SUMMARY:
This study aimed to evaluate the anticancer activity of capmatinib in combination with osimertinib compared to platinum-pemetrexed based doublet chemotherapy as second line treatment in patients with advanced or metastatic non-small-cell lung cancer (NSCLC) with epidermal growth factor receptor (EGFR) mutation, T790M negative, mesenchymal-to-epithelial transition factor (MET) amplified who progressed following EGFR tyrosine kinase inhibitors (TKIs).

DETAILED DESCRIPTION:
This was a multicenter, open-label, randomized, active-controlled, global phase III study that enrolled adult participants with locally advanced or metastatic NSCLC with epidermal growth factor receptor (EGFR) activating mutation, T790M negative, mesenchymal-to-epithelial transition factor (MET) amplified who had progressed following EGFR tyrosine kinase inhibitors (TKIs).

The study was conducted in two parts. The initial part was a safety run-in part, which aimed at assessing the safety and tolerability of capmatinib in combination with osimertinib and at determining the recommended dosage for the subsequent randomized part. The randomized part compared the efficacy and safety of capmatinib in combination with osimertinib to a platinum-based doublet chemotherapy regimen using either cisplatin or carboplatin, combined with pemetrexed, as second-line treatment.The randomized part was not initiated.

In the randomized part (if initiated), participants were to receive their assigned treatment (either capmatinib in combination with osimertinib or platinum-pemetrexed based doublet chemotherapy) until they experienced any of the following: documented disease progression according to the Response Evaluation Criteria In Solid Tumors 1.1 (RECIST 1.1) as assessed by the investigator during the run-in part and confirmed by a blinded independent review committee (BIRC) during the randomized part, withdrawal of consent, pregnancy, lost to follow-up, or death. Participants who progressed in the platinum-pemetrexed arm were to be permitted to switch to capmatinib in combination with osimertinib therapy after BIRC-confirmed, RECIST 1.1-defined progressive disease. If, in the judgment of the investigator, there was evidence of clinical benefit and the participant wished to continue, study treatment could be continued beyond the initial disease progression according to RECIST 1.1 criteria. After treatment discontinuation, all participants were to be followed for safety evaluations during the safety follow-up period.

On 11-May-2022, Novartis decided to halt enrollment for this study due to a business consideration unrelated to any safety concerns. Ongoing patients in the run-in part were allowed to continue treatment through other post-trial drug supply options, as applicable. On 27-Dec-2022 the last patient was transitioned off the study, and following the study protocol this date was declared the Global end of trial date. Randomized part was not initiated.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of NSCLC with EGFR mutations known to be associated with EGFR TKI sensitivity, EGFR T790M negative and MET gene amplification
* Stage IIIB/IIIC or IV NSCLC
* Participants must have progressed on one prior line of therapy (1st/2nd generation EGFR TKIs, osimertinib or other third generation EGFR TKIs) for advanced/metastatic disease (stage IIIB/IIIC and must be candidates for platinum (cisplatin or carboplatin) - pemetrexed doublet based chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Participants must have recovered from all toxicities related to prior systemic therapy to grade ≤ 1 Common Terminology Criteria Adverse Event 5.0 (CTCAE v 5.0)
* At least one measurable lesion as defined by RECIST 1.1
* Participants must have adequate organ function

Key Exclusion Criteria:

* Prior treatment with any MET inhibitor or HGF-targeting therapy
* Participants with symptomatic central nervous system (CNS) metastases who were neurologically unstable or had required increasing doses of steroids within the 2 weeks prior to study entry to manage CNS symptoms
* Carcinomatous meningitis
* Presence or history of a malignant disease other than NSCLC that had been diagnosed and/or required therapy within the past 3 years
* Presence or history of interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis
* Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome
* Clinically significant, uncontrolled heart diseases
* known druggable molecular alterations that may render participants eligible for alternative targeted therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Japan (2):
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Sunto Gun, Shizuoka
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- See also: Plain Language Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1727

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In the run-in part, participants were enrolled at 4 investigative sites in 3 countries. The study was terminated early based on Sponsor's decision unrelated to any safety concerns and the randomized part of the study was not initiated.
Pre-assignment Details: A total of 23 participants were screened of which 6 participants were enrolled into the run-in part of the study.
Groups:
- Run-in Part: Capmatinib + Osimertinib: Participants received a starting dose of capmatinib 400 mg, orally, twice daily (BID) in combination with osimertinib 80 mg, orally, once daily (QD)
Period: Overall Study
Arm/Group | Run-in Part: Capmatinib + Osimertinib | Randomized Part: Capmatinib + Osimertinib | Randomized Part: Platinum + Pemetrexed Based Doublet Chemotherapy
Started | 6 | 0 | 0
Full Analysis Set (FAS) (FAS included all participants who received any component of the study treatment.) | 6 | 0 | 0
Safety Set (Safety set included all participants who received at least one dose of study treatment.) | 6 | 0 | 0
Pharmacokinetic (PK) Analysis Set (PK analysis set included all participants who provided at least one evaluable PK concentration.) | 6 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 6 | 0 | 0
Not completed — Progressive Disease | 4 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Study Terminated by Sponsor | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Run-in Part: Capmatinib + Osimertinib
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (7.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Run-in Part: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: A DLT was defined as an adverse event (AE) or abnormal laboratory value assessed as unrelated to disease, progressive disease, inter-current illness, or concomitant medications, that despite optimal therapeutic intervention that occurred within the first 21 days of treatment with capmatinib in combination with osimertinib.
Time Frame: Up to 21 Days
Population: FAS included all participants who received any component of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Part: Capmatinib + Osimertinib
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: Randomized Part: Progression Free Survival (PFS) Based on BIRC Assessment
Description: PFS was defined as time from date of randomization to the date of first documented disease progression (PD) based on Blinded Independent Review Committee (BIRC) as per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1), or death from any cause, whichever occurred first. Progression was defined as a ≥20% increase in sum of longest diameters (SLD) compared to smallest SLD in the study, or progression of non-target lesions or new lesions.
Time Frame: From randomization to first documented progression or deaths, planned to be assessed up to 37 months
Population: Due to early study termination, the randomized part of the study was not initiated. Hence the data was not collected for the outcome measures in the randomized part of the study.
Arm/Group | Randomized Part: Capmatinib + Osimertinib | Randomized Part: Platinum + Pemetrexed Based Doublet Chemotherapy
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Run-in Part: Number of Participants With at Least One Dose Interruption and Dose Reduction of Each Study Drug
Description: Number of participants with at least one dose interruption and dose reduction were reported for each study drug.
Time Frame: From the first dose until last dose of study treatment, assessed up to 39 weeks
Population: Safety set included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Part: Capmatinib + Osimertinib
Number analyzed (Participants) | 6
Participants
  Dose Interruption: Capmatinib | 5
  Dose Interruption: Osimertinib | 4
  Dose Reduction: Capmatinib | 3
  Dose Reduction: Osimertinib | 0

4. Secondary Outcome: Run-in Part: Dose Intensity of Each Study Drug
Description: Dose intensity was computed as the ratio of actual cumulative dose (milligrams) received and actual duration of exposure (weeks) to study drug.
Time Frame: From the first dose until last dose of study treatment, assessed up to 39 weeks
Population: Safety set included all participants who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: milligrams per week (mg/week)
Arm/Group | Run-in Part: Capmatinib + Osimertinib
Number analyzed (Participants) | 6
milligrams per week (mg/week)
  Capmatinib | 5042.8 (947.28)
  Osimertinib | 534.9 (41.29)

5. Secondary Outcome: Run-in Part: Median Duration of Exposure to Each Study Drug
Description: Duration of exposure is defined as the time (in weeks) between the first and the last dose of study treatment.
Time Frame: From the first dose until last dose of study treatment, assessed up to 39 weeks
Population: Safety set included all participants who received at least one dose of study treatment.
Measure: Median (Full Range); unit: weeks
Arm/Group | Run-in Part: Capmatinib + Osimertinib
Number analyzed (Participants) | 6
weeks
  Capmatinib | 23.5 [1 to 39]
  Osimertinib | 24.0 [1 to 39]

6. Secondary Outcome: Run-in Part: Maximum Plasma Concentration (Cmax) of Capmatinib
Description: Blood samples were collected. Cmax of capmatinib was calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
  Actual recorded sampling times were considered for the calculations
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, and 8 hours post-dose on Days 1 and 15 of Cycle 1 (Cycle = 21 days)
Population: PK analysis set included all participants who provided at least one evaluable PK concentration. 'Number analyzed' indicates the number of participants with data available for analysis at specified timepoint.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Run-in Part: Capmatinib + Osimertinib
Number analyzed (Participants) | 6
nanograms per milliliter (ng/mL)
  Day 1 | 5510 (2380)
  Day 15: number analyzed (Participants) | 5
  Day 15 | 5750 (1050)

7. Secondary Outcome: Run-in Part: Maximum Plasma Concentration (Cmax) of Osimertinib and Its Metabolites (AZ5104 and AZ7550)
Description: Blood samples were collected. Cmax of osimertinib and its metabolites (AZ5104 and AZ7550) was calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8 and 24 hours post-dose on Days 1 and 15 of Cycle 1 (Cycle = 21 days)
Population: PK analysis set included all participants who provided at least one evaluable PK concentration. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis. 'Number analyzed' indicates the number of participants with data available at specified timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Run-in Part: Capmatinib + Osimertinib
Number analyzed (Participants) | 5
ng/mL
  Osimertinib: Day 1 | 99.5 (57.0)
  Osimertinib: Day 15 | 265 (113)
  AZ5104: Day 1 | 4.86 (3.22)
  AZ5104: Day 15 | 22.0 (9.23)
  AZ7550: Day 1 | 3.61 (1.53)
  AZ7550: Day 15: number analyzed (Participants) | 4
  AZ7550: Day 15 | 33.0 (11.9)

8. Secondary Outcome: Run-in Part: Time to Maximum Plasma Concentration (Tmax) of Capmatinib
Description: Blood samples were collected. Tmax of capmatinib was calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
  Actual recorded sampling times were considered for the calculations
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, and 8 hours post-dose on Days 1 and 15 of Cycle 1 (Cycle = 21 days)
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | Run-in Part: Capmatinib + Osimertinib
Number analyzed (Participants) | 6
hours
  Day 1 | 1.92 [0.983 to 3.02]
  Day 15: number analyzed (Participants) | 5
  Day 15 | 1.00 [0.917 to 1.82]

9. Secondary Outcome: Run-in Part: Time to Maximum Plasma Concentration (Tmax) of Osimertinib and Its Metabolites (AZ5104 and AZ7550)
Description: Blood samples were collected. Tmax of osimertinib and its metabolites (AZ5104 and AZ7550) was calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
  Actual recorded sampling times were considered for the calculations
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8 and 24 hours post-dose on Days 1 and 15 of Cycle 1 (Cycle = 21 days)
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Run-in Part: Capmatinib + Osimertinib
Number analyzed (Participants) | 5
hours
  Osimertinib: Day 1 | 6.00 [2.90 to 23.1]
  Osimertinib: Day 15 | 4.00 [0.00 to 7.33]
  AZ5104: Day 1 | 23.1 [22.3 to 23.5]
  AZ5104: Day 15 | 4.00 [0.00 to 7.13]
  AZ7550: Day 1 | 5.68 [2.90 to 23.1]
  AZ7550: Day 15: number analyzed (Participants) | 4
  AZ7550: Day 15 | 2.25 [0.00 to 6.00]

10. Secondary Outcome: Run-in Part: Area Under the Curve to the Last Measurable Concentration (AUClast) of Capmatinib
Description: Blood samples were collected. AUClast of capmatinib was calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, and 8 hours post-dose on Days 1 and 15 of Cycle 1 (Cycle = 21 days)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: nanograms*hours/milliliter (ng*hr/mL)
Arm/Group | Run-in Part: Capmatinib + Osimertinib
Number analyzed (Participants) | 6
nanograms*hours/milliliter (ng*hr/mL)
  Day 1 | 20100 (6080)
  Day 15: number analyzed (Participants) | 5
  Day 15 | 21300 (7050)

11. Secondary Outcome: Run-in Part: Area Under the Curve to the Last Measurable Concentration (AUClast) of Osimertinib and Its Metabolites (AZ5104 and AZ7550)
Description: Blood samples were collected. AUClast of osimertinib and its metabolites (AZ5104 and AZ7550) was calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8 and 24 hours post-dose on Days 1 and 15 of Cycle 1 (Cycle = 21 days)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Run-in Part: Capmatinib + Osimertinib
Number analyzed (Participants) | 5
ng*hr/mL
  Osimertinib: Day 1 | 1790 (1030)
  Osimertinib: Day 15 | 1380 (900)
  AZ5104: Day 1 | 82.9 (59.4)
  AZ5104: Day 15 | 136 (56.8)
  AZ7550: Day 1 | 47.1 (46.3)
  AZ7550: Day 15: number analyzed (Participants) | 4
  AZ7550: Day 15 | 112 (111)

12. Secondary Outcome: Run-in Part: Overall Response Rate (ORR) as Per Investigator Assessment
Description: ORR was defined as the percentage of participants with a confirmed best overall response (BOR) of complete response (CR) or partial response (PR), as per investigator judgment and according to RECIST v1.1. Criteria for CR: Disappearance of all lesions and pathologic lymph nodes; PR: ≥30% decrease in the SLD of the target lesions or no new lesions or no progression of non-target lesions.
Time Frame: Up to end of study, assessed up to 39 weeks
Population: FAS included all participants who received any component of the study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Run-in Part: Capmatinib + Osimertinib
Number analyzed (Participants) | 6
percentage of participants | 50.0 [11.8 to 88.2]

13. Secondary Outcome: Run-in Part: Duration of Response (DOR) as Per Investigator Assessment
Description: DOR was defined as the time from first documented response of CR or PR to the date of first documented PD or death due to any cause. Criteria for CR: Disappearance of all lesions and pathologic lymph nodes; PR: ≥30% decrease in the SLD of the target lesions or no new lesions or no progression of non-target lesions; PD: ≥20% increase in SLD compared to the smallest SLD in the study, or progression of non-target lesions or new lesions.
Time Frame: Up to disease progression or death or end of study, assessed up to 39 weeks
Population: FAS included all participants who received any component of the study treatment. 'Overall number of participants analyzed' indicates the number of participants with CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Run-in Part: Capmatinib + Osimertinib
Number analyzed (Participants) | 3
months | 6.93 [2.50 to NA] — Upper limit of 95% confidence interval (CI) was not estimable due to an insufficient number of participants with events.

14. Secondary Outcome: Run-in Part: Time to Response (TTR) as Per Investigator Assessment
Description: TTR was defined as the duration of time between the date of fist dose of treatmwnr and the date of the first documented response of either CR or PR as per investigator judgment and according to RECIST v1.1 criteria. Criteria for CR: Disappearance of all lesions and pathologic lymph nodes; PR: ≥30% decrease in SLD of the target lesions or no new lesions or no progression of non-target lesions.
Time Frame: From first dose of treatment up to end of study, assessed up to 39 weeks
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Run-in Part: Capmatinib + Osimertinib
Number analyzed (Participants) | 3
months | NA [1.41 to NA] — Median and the upper limit of 95% CI were not estimable due to an insufficient number of participants with events.

15. Secondary Outcome: Run-in Part: Disease Control Rate (DCR) as Per Investigator Assessment
Description: DCR was defined as the percentage of participants with a BOR of CR, PR, and stable disease (SD) as per investigator judgment and according to RECIST v1.1. Criteria for CR: Disappearance of all lesions and pathologic lymph nodes; PR: ≥30% decrease in SLD of the target lesions or no new lesions or no progression of non-target lesions; SD: Neither sufficient shrinkage to qualify for PR or CR nor and increase in lesions which would qualify for PD. PD: ≥20% increase in SLD compared to the smallest SLD in the study, or progression of non-target lesions or new lesions.
Time Frame: From randomization up to end of study, assessed up to 39 weeks
Population: FAS included all participants who received any component of the study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Run-in Part: Capmatinib + Osimertinib
Number analyzed (Participants) | 6
percentage of participants | 66.7 [22.3 to 95.7]

16. Secondary Outcome: Run-in Part: Progression-Free Survival (PFS) as Per Investigator Assessment
Description: PFS was defined as the time (in months) from first dose of treatment to the date of the first documented progression or death due to any cause as per investigator judgment and according to RECIST v1.1. Progression was defined as a ≥20% increase in SLD compared to smallest SLD in the study, or progression of non-target lesions or new lesions. PFS was censored if no PFS event (progression or death) was observed.
Time Frame: From first dose of treatment until first documented progression or death or end of study, assessed up to 39 weeks
Population: FAS included all participants who received any component of the study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Run-in Part: Capmatinib + Osimertinib
Number analyzed (Participants) | 6
months | 4.58 [0.99 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with events.

17. Secondary Outcome: Randomized Part: Overall Response Rate (ORR) as Per BIRC Assessment
Description: ORR was defined as the percentage of participants with confirmed BOR of CR or PR, as per BIRC by RECIST v1.1. Criteria for CR: Disappearance of all lesions and pathologic lymph nodes; PR: ≥30% decrease in SLD of the target lesions or no new lesions or no progression of non-target lesions.
Time Frame: Planned to be assessed up to 37 months
Population: Due to early study termination, the randomized part of the study was not conducted. Hence the data was not collected for the outcome measures in the randomized part of the study.
Arm/Group | Randomized Part: Capmatinib + Osimertinib | Randomized Part: Platinum + Pemetrexed Based Doublet Chemotherapy
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Randomized Part: Overall Intracranial Response Rate (OIRR) as Per BIRC Assessment
Description: OIRR was defined as the percentage of participants with a confirmed best overall intracranial response (BOIR) of CR or PR as per BIRC according to Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria. Criteria for CR: Disappearance of all CNS target and non-target lesions sustained for at least 4 weeks, with no new lesions, and no use of corticosteroids. PR: ≥30% decrease in the SLD of CNS target lesions or no new lesions or and stable to decreased corticosteroid dose.
Time Frame: Planned to be assessed up to 37 months
Population: as for outcome 17
Arm/Group | Randomized Part: Capmatinib + Osimertinib | Randomized Part: Platinum + Pemetrexed Based Doublet Chemotherapy
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Randomized Part: Duration of Response (DOR) as Per BIRC Assessment
Description: DOR was defined as the time from the first documented response of CR or PR to the date of first documented progression or death as per BIRC according to RECIST v1.1 criteria. Criteria for CR: Disappearance of all lesions and pathologic lymph nodes; PR: ≥30% decrease in SLD of the target lesions or no new lesions or no progression of non-target lesions; PD: ≥20% increase in SLD compared to the smallest SLD in the study, or progression of non-target lesions or new lesions.
Time Frame: From first documented response to first documented progression or death, planned to be assessed up to 37 months
Population: as for outcome 17
Arm/Group | Randomized Part: Capmatinib + Osimertinib | Randomized Part: Platinum + Pemetrexed Based Doublet Chemotherapy
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Randomized Part: Time to Response (TTR) as Per BIRC Assessment
Description: TTR was defined as duration of time between the date of randomization and the date of first documented response of either CR or PR as per BIRC according to RECIST v1.1 criteria. Criteria for CR: Disappearance of all lesions and pathologic lymph nodes; PR: ≥30% decrease in SLD of the target lesions or no new lesions or no progression of non-target lesions.
Time Frame: From randomization to first documented response, planned to be assessed up to 37 months
Population: as for outcome 17
Arm/Group | Randomized Part: Capmatinib + Osimertinib | Randomized Part: Platinum + Pemetrexed Based Doublet Chemotherapy
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Randomized Part: Disease Control Rate (DCR) as Per BIRC Assessment
Description: DCR was defined as the percentage of participants with CR or PR or SD as per BIRC according to RECIST v1.1 criteria. Criteria for CR: Disappearance of all lesions and pathologic lymph nodes; PR: ≥30% decrease in SLD of the target lesions or no new lesions or no progression of non-target lesions; SD: Neither sufficient shrinkage to qualify for PR or CR nor and increase in lesions which would qualify for PD. PD: ≥20% increase in SLD compared to the smallest SLD in the study, or progression of non-target lesions or new lesions.
Time Frame: Planned to be assessed up to 37 months
Population: as for outcome 17
Arm/Group | Randomized Part: Capmatinib + Osimertinib | Randomized Part: Platinum + Pemetrexed Based Doublet Chemotherapy
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Randomized Part: Progression-Free Survival After Next Line of Treatment (PFS2) as Per Investigator Assessment
Description: PFS2 was defined as the time from date of randomization to the first documented progression on the next line therapy as per investigator judgment according to RECIST v1.1 response criteria or death due to any cause.
Time Frame: Planned to be assessed up to 37 months
Population: as for outcome 17
Arm/Group | Randomized Part: Capmatinib + Osimertinib | Randomized Part: Platinum + Pemetrexed Based Doublet Chemotherapy
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Randomized Part: Maximum Plasma Concentration (Cmax) of Capmatinib
Description: Cmax of capmatinib calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Time Frame: Pre-dose on Day 1 of Cycles 1, 2, 3, 4 and 6 (Cycle = 21 days)
Population: as for outcome 17
Arm/Group | Randomized Part: Capmatinib + Osimertinib | Randomized Part: Platinum + Pemetrexed Based Doublet Chemotherapy
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Randomized Part: Maximum Plasma Concentration (Cmax) of Osimertinib and Its Metabolites
Description: Cmax of osimertinib and its metabolites (AZ5104 and AZ7550) calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Time Frame: Pre-dose on Day 1 of Cycles 1, 2, 3, 4 and 6 (Cycle = 21 days)
Population: as for outcome 17
Arm/Group | Randomized Part: Capmatinib + Osimertinib | Randomized Part: Platinum + Pemetrexed Based Doublet Chemotherapy
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Randomized Part: Overall Survival (OS)
Description: OS was defined as the time from date of randomization to date of death due to any cause.
Time Frame: From randomization to date of death, planned to be assessed up to 37 months
Population: as for outcome 17
Arm/Group | Randomized Part: Capmatinib + Osimertinib | Randomized Part: Platinum + Pemetrexed Based Doublet Chemotherapy
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Randomized Part: Change From Baseline in the European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life Questionnaire (EORTC QLQ-C30) Score
Description: EORTC QLQ-C30 is a questionnaire developed to assess the quality of life of cancer patients. It contains 30 items and is composed of both multi-item scales and single-item measures based on the participant's experience over the past week. These include five scales (physical, role, emotional, cognitive, and social functioning), three symptom scales (fatigue, nausea/vomiting, and pain), six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial impact) and a global health status/quality of life scale (QoL) scale. All of the scales and single-item measures range in score from 0 to 100. A high score for a functional scale represents a high /healthy level of functioning; a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology/problems.
Time Frame: Cycle 1 Day 1, Cycle 3 Day 1, then every 6 weeks for the 18 months after Cycle 1 Day 1 and every 12 weeks thereafter, until end of treatment, end of treatment and 6, 12 and 18 weeks post-progression (Cycle = 21 days)
Population: as for outcome 17
Arm/Group | Randomized Part: Capmatinib + Osimertinib | Randomized Part: Platinum + Pemetrexed Based Doublet Chemotherapy
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Randomized Part: Change From Baseline in the EORTC QLQ Lung Cancer Module (EORTC QLQ-LC13) Score
Description: EORTC QLQ-LC13 is used in conjunction with the EORTC QLQ-C30 and provides information on an additional 13 items specifically related to lung cancer. The five domains of the LC13 include pain, dyspnea, coughing and hemoptysis, and are based on their presence over the past week. All but the pain domain are scored on a 4 point Likert scale ranging from "not at all" to "very much". Pain score is based on its presence, hence yes or no. Scores are averaged and transformed to 0 to 100. A higher score indicates a higher presence of symptoms.
Time Frame: as for outcome 26
Population: as for outcome 17
Arm/Group | Randomized Part: Capmatinib + Osimertinib | Randomized Part: Platinum + Pemetrexed Based Doublet Chemotherapy
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Randomized Part: Change From Baseline in the EuroQoL-5 Dimension-5 Level (EQ-5D-5L) Score
Description: EQ-5D-5L is a standardized measure of health status developed by the EuroQol (EQ) Group in order to provide a simple, generic measure of health for clinical and economic appraisal. The EQ-5D-5L consists of 2 pages - the descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). For each of these dimensions, the participant self-assigned a score: from 1 (no problems) to 5 (extreme problems). The questionnaire also includes a Visual Analogue Scale (VAS), where the participant is asked to rate current health status on a scale of 0 to 100, with 0 being the worst imaginable health state.
Time Frame: as for outcome 26
Population: as for outcome 17
Arm/Group | Randomized Part: Capmatinib + Osimertinib | Randomized Part: Platinum + Pemetrexed Based Doublet Chemotherapy
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Randomized Part: Change From Baseline in the National Comprehensive Cancer Network Functional Assessment of Cancer Therapy (NCCN FACT)-Brain Symptom Index Version 2.0 (FBrSI)
Description: The NCCN FACT-Brain Symptom Index version 2.0 (FBrSI) is a questionnaire used to explore changes in symptoms associated with potential brain metastases (BM). The symptoms module contains 12 items with a recall period of the past 7 days. The participant responds to 12 statements and indicates to what extent it applies to them on a 5-point Likert response scale from "not at all"=0 to "very much"=4. Higher scores indicates a greater impact of symptoms on the participant's quality of life.
Time Frame: as for outcome 26
Population: as for outcome 17
Arm/Group | Randomized Part: Capmatinib + Osimertinib | Randomized Part: Platinum + Pemetrexed Based Doublet Chemotherapy
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Randomized Part: Time to Symptom Deterioration for EORTC QLQ-C30 Questionnaire
Description: Time to symptom deterioration from baseline from baseline for participant scores from the EORTC QLQ-C30 questionnaire. EORTC QLQ-C30 is a questionnaire developed to assess the quality of life of cancer patients. It contains 30 items and is composed of both multi-item scales and single-item measures based on the participant's experience over the past week. These include five scales (physical, role, emotional, cognitive, and social functioning), three symptom scales (fatigue, nausea/vomiting, and pain), six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial impact) and a global health status/quality of life scale (QoL) scale. All of the scales and single-item measures range in score from 0 to 100. A high score for a functional scale represents a high /healthy level of functioning; a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology/problems.
Time Frame: From baseline to symptom deterioration, planned to be assessed up to 37 months
Population: as for outcome 17
Arm/Group | Randomized Part: Capmatinib + Osimertinib | Randomized Part: Platinum + Pemetrexed Based Doublet Chemotherapy
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Randomized Part: Time to Symptom Deterioration for EORTC QLQ-LC13 Questionnaire
Description: Time to symptom deterioration from baseline for participant scores from EORTC QLQ-LC13 questionnaire. EORTC QLQ-LC13 is used in conjunction with the EORTC QLQ-C30 and provides information on an additional 13 items specifically related to lung cancer. The five domains of the LC13 include pain, dyspnea, coughing and hemoptysis, and are based on their presence over the past week. All but the pain domain are scored on a 4 point Likert scale ranging from "not at all" to "very much". Pain score is based on its presence, hence yes or no. Scores are averaged and transformed to 0 to 100. A higher score indicates a higher presence of symptoms.
Time Frame: From baseline to symptom deterioration, planned to be assessed up to 37 months
Population: as for outcome 17
Arm/Group | Randomized Part: Capmatinib + Osimertinib | Randomized Part: Platinum + Pemetrexed Based Doublet Chemotherapy
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: Randomized Part: Time to Symptom Deterioration for NCCN FBrSl Questionnaire
Description: Time to symptom deterioration from baseline for participant scores from the NCCN FBrSl questionnaire. The NCCN FACT-Brain Symptom Index version 2.0 (FBrSI) is a questionnaire used to explore changes in symptoms associated with potential brain metastases (BM). The symptoms module contains 12 items with a recall period of the past 7 days. The participant responds to 12 statements and indicates to what extent it applies to them on a 5-point Likert response scale from "not at all"=0 to "very much"=4. Higher scores indicates a greater impact of symptoms on the participant's quality of life.
Time Frame: From baseline to symptom deterioration, planned to be assessed up to 37 months
Population: as for outcome 17
Arm/Group | Randomized Part: Capmatinib + Osimertinib | Randomized Part: Platinum + Pemetrexed Based Doublet Chemotherapy
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: Randomized Part: Duration of Intracranial Response (DOIR) Based on BIRC
Description: DOIR was defined as the time from the date of first documented intracranial response of either CR or PR to the date of the first documented intracranial progression per RANO-BM criteria as assessed by BIRC review or the date of death due to any cause. Criteria for CR: Disappearance of all CNS target and non-target lesions sustained for at least 4 weeks, with no new lesions, and no use of corticosteroids; PR: ≥30% decrease in the SLD of CNS target lesions or no new lesions, and stable to decreased corticosteroid dose.
Time Frame: From the date of first documented intracranial response to first documented intracranial progression or death, planned to be assessed up to 37 months
Population: as for outcome 17
Arm/Group | Randomized Part: Capmatinib + Osimertinib | Randomized Part: Platinum + Pemetrexed Based Doublet Chemotherapy
Number analyzed (Participants) | 0 | 0

34. Secondary Outcome: Randomized Part: Time to Intracranial Response (TTIR) Based on BIRC
Description: TTIR was defined as the time from the date of randomization to the date of the first documented intracranial response of either CR or PR as per BIRC according to RANO-BM criteria. Criteria for CR: Disappearance of all CNS target and non-target lesions sustained for at least 4 weeks, with no new lesions, and no use of corticosteroids; PR: ≥30% decrease in the SLD of CNS target lesions or no new lesions, and stable to decreased corticosteroid dose.
Time Frame: From randomization to first documented response, planned to be assessed up to 37 months
Population: as for outcome 17
Arm/Group | Randomized Part: Capmatinib + Osimertinib | Randomized Part: Platinum + Pemetrexed Based Doublet Chemotherapy
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: Randomized Part: Intracranial Disease Control Rate (IDCR) Based on BIRC
Description: IDCR was defined as the percentage of participants with a confirmed BOIR of CR or PR or SD as per BIRC according to RANO-BM criteria. Criteria for CR: Disappearance of all CNS target and non-target lesions sustained for at least 4 weeks, with no new lesions, and no use of corticosteroids; PR: ≥30% decrease in the SLD of CNS target lesions or no new lesions, and stable to decreased corticosteroid dose; SD: Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease.
Time Frame: Planned to be assessed up to 37 months
Population: as for outcome 17
Arm/Group | Randomized Part: Capmatinib + Osimertinib | Randomized Part: Platinum + Pemetrexed Based Doublet Chemotherapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of treatment until 30 days after last dose of study treatment, assessed up to 39 weeks.
Description: Safety set included all participants who received at least one dose of study treatment. Due to early study termination, the randomized part of the study was not conducted. Hence safety data was not collected in the randomized part of the study.
Arm/Group | Run-in Part: Capmatinib + Osimertinib
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Part: Capmatinib + Osimertinib (N=6)
Pericardial effusion (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 1
COVID-19 (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Part: Capmatinib + Osimertinib (N=6)
Neutropenia (Blood and lymphatic system disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 1
Cataract (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 1
Oedema peripheral (General disorders) | 4
Peripheral swelling (General disorders) | 1
Pyrexia (General disorders) | 1
COVID-19 (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Amylase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Lipase increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/14/NCT04816214/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/14/NCT04816214/SAP_001.pdf